CLINICAL TRIAL: NCT01951820
Title: Comparison of Efficacy of Two Topical Anesthetics: Benzocaine Versus Pliaglis for Control of Pain Associated With Dental Needle Insertion in the Palate, A Double Blind Study
Brief Title: Comparison of Two Topical Anesthetics: Benzocaine Versus Pliaglis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Association of Endodontists (Other)
Responsible Party: Principal Investigator, Brian Royle, Endodontic Resident, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUM00075036
Record Dates: First submitted 2013-08-22; First posted 2013-09-27 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia of Mucous Membrane
MeSH Terms: interventions — Lidocaine; Tetracaine; Benzocaine; Carticaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benzocaine (Active Comparator): Benzocaine topical numbing gel will be applied to the gums before injection with other intervention, injection of local anesthetic articaine.
  Interventions: Drug: Benzocaine; Drug: Articaine
- Pliaglis (Experimental): Pliaglis topical numbing gel will be applied to the gums before injection with other intervention, injection of local anesthetic articaine.
  Interventions: Drug: Pliaglis; Drug: Articaine

INTERVENTIONS:
Drug: Pliaglis — Apply 0.2mg of compounded topical anesthetic (Pliaglis) to gums for 2.5 minutes before giving patient injection of local anesthetic.
  Other Names: lidocaine and tetracaine
  Arms: Pliaglis
Drug: Benzocaine — Apply 0.2mg of topical anesthetic (benzocaine) to gums for 2.5 minutes before giving patient injection of local anesthetic.
  Other Names: Hurricaine
  Arms: Benzocaine
Drug: Articaine — Injection of 0.4mg of local anesthetic in gum tissue where topical anesthetic was placed
  Other Names: Septocaine

SUMMARY:
The efficacy of the topical anesthetics will be determined by how much pain the patient felt (using a Heft-Parker pain analog scale) upon needle penetration.

DETAILED DESCRIPTION:
This project will be a double blind study comparing the efficacy of two different topical anesthetics used to reduce the pain associated with insertion of dental needles on the palatal mucosa. The two topical anesthetics being compared are 20% Benzocaine, and Pliaglis.

In order to complete a number of different dental procedures, it is often necessary to provide local anesthesia of the palate. Intraoral injections into the palatal mucosa are often uncomfortable and even painful. In an effort to increase patient comfort, a topical anesthetic is often used prior to the injection. Test subjects undergoing routine endodontic treatment on maxillary teeth will have a 27- gauge dental needle inserted into the mucosa of the hard palate as part of the initial step in standard local anesthetic injection. At the injection site and prior to the needle stick, the mucosa will be topically anesthetized by using one of the two different test compounds (Benzocaine or Pliaglis). After the injection, patients will be asked to score the level of discomfort associated with the needle stick.

The purpose of the project is to determine if there is a clinical difference in the level of pain felt upon needle stick, between the two different topical anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* normal healthy adults 18+ yrs old requiring root canal treatment of maxillary molars
* Patients with healthy mucosal tissues, and who do not have pain on palpation at injection site
* Ability to use and understand a VAS score
* Ability to use and understand a VAS score
* No know allergies to topical anesthetics being used

Exclusion Criteria:

* Allergy or other contraindications to topical anesthetics
* Allergy to epinephrine or local anesthetics
* Broken/unhealthy mucosal tissues and pain on palpation at injection site
* Patients needing endodontic therapy on maxillary anterior teeth
* Inability to consent to participate in the study
* Patients who have used analgesics within 6 hours of appointment time
* Pregnant and nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian l Royle, DDS, Principal Investigator — University of Michigan department of Endodontics
Locations (1):
- University of Michigan Dental School, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Benzocaine | Pliaglis
Started | 34 | 30
Completed | 34 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benzocaine | Pliaglis | Total
Number analyzed (Participants) | 34 | 30 | 64
Age, Customized [Number; unit: participants]
  >18 Years | 34 | 30 | 64
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 17 | 15 | 32
Region of Enrollment [Number; unit: participants]
  United States | 34 | 30 | 64

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Pain Associated With Injection, in Millimeters, According to Visual Analog Scale
Description: The investigation is trying to determine if the compounded topical anesthetic (Pliaglis) is more effective than the active control (benzocaine) in numbing the gums before needle penetration. The effectiveness of the topical anesthetics will be determined by the patient indicating their level of discomfort felt upon needle stick by using a Heft-Parker visual analog pain scale (scale of 0 - 170mm with 0mm equating to no pain and 170mm equating to maximum pain).
Time Frame: 2.5 minutes
Measure: Mean (Full Range); unit: mm
Arm/Group | Benzocaine | Pliaglis
Number analyzed (Participants) | 34 | 30
mm | 38.5 [0 to 170] | 26.9 [0 to 170]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Benzocaine | Pliaglis
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/30
Other Adverse Events (participants affected / at risk) | 0/34 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No